CLINICAL TRIAL: NCT07074938
Title: A Non-inferiority Randomized Controlled Study Comparing Jianmin Daopeng An Gong Niuhuang Wan and Tongrentang An Gong Niuhuang Wan in Promoting the Postoperative Neurological Function Recovery of Patients With Traumatic Brain Injury
Brief Title: An Gong Niuhuang Wan Promotes the Postoperative Neurological Function Recovery of Patients With Traumatic Brain Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huaqiu Zhang (Other)
Responsible Party: Sponsor-Investigator, Huaqiu Zhang, Clinical Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TJ-IRB202504084
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jianmin Dapeng Angong Niuhuang Wan (Experimental): Jianmin Dapeng Angong Niuhuang Wan. All the enrolled patients were given oral medication. For those who were unable to eat independently, nasogastric administration was carried out using warm water to dissolve the medicine. Usage and dosage: Oral administration, 1 pill each time, once a day, for 1 week.
  Interventions: Drug: Jianmin Daopeng Angong Niuhuang Wan
- Tongrentang Angong Niuhuang Wan (Sham Comparator): Tongrentang Angong Niuhuang Wan. All the enrolled patients were given oral medication. For those who were unable to eat independently, nasogastric administration was carried out using warm water to dissolve the medicine. Usage and dosage: Oral administration, 1 pill each time, once a day, for 1 week.
  Interventions: Drug: Tongrentang Angong Niuhuang Wan

INTERVENTIONS:
Drug: Jianmin Daopeng Angong Niuhuang Wan — An Gong Niu Huang Wan comes from JianMin Dapeng.
  Arms: Jianmin Dapeng Angong Niuhuang Wan
Drug: Tongrentang Angong Niuhuang Wan — Angong Niuhuang Wan comes from Tongrentang.
  Arms: Tongrentang Angong Niuhuang Wan

SUMMARY:
Clinical Challenges and Severity of Traumatic Brain Injury: Traumatic brain injury, as a common neurosurgical disease, poses a significant threat to patients' life safety and quality of life.The promotion of in vitro cultivated cow bile in the treatment of post-traumatic brain injury is expected to provide a more economical and effective treatment option for the recovery of consciousness and cognitive functions of TBI patients. Compared with traditional An Gong Niu Huang Wan, Jian Min Da Peng's An Gong Niu Huang Wan (containing in vitro cultivated cow bile) can not only reduce treatment costs, but also improve the stability and consistency of the quality of the drug. The above clinical research can provide scientific basis for including it in relevant treatment guidelines.

DETAILED DESCRIPTION:
Clinical Challenges and Severity of Traumatic Brain Injury: Traumatic brain injury, as a common neurosurgical disease, poses a significant threat to patients' life safety and quality of life. Post-operative patients with traumatic brain injury often suffer from severe neurological impairments, consciousness disorders, systemic inflammatory responses, and even pose a threat to their lives. The recovery of consciousness and cognitive functions is of great significance for patients' quality of life and functional rehabilitation.

Clinical Status: Currently, the treatment methods for traumatic brain injury include early emergency surgical treatment of the primary injury (such as surgical removal of intracranial hematoma, contusion and laceration of brain tissue, etc.) and post-operative drug and rehabilitation treatment for secondary neurological dysfunction (including but not limited to neurological function recovery, treatment of brain tissue edema, treatment of cerebral ischemia and its systemic inflammatory responses). For a long time, An Gong Niu Huang Wan has been used as a traditional Chinese medicine for some patients with clinical brain injury due to its significant pharmacological functions such as anti-inflammatory and clearing heat, awakening the mind and opening the orifices. However, due to the scarcity and high price of the active ingredient "natural cow bile" in An Gong Niu Huang Wan, its wide application in these patients has been limited. Jian Min Da Peng An Gong Niu Huang Wan is a kind of artificial cow bile synthesized and cultivated in the laboratory through in vitro cultivation, which has similar pharmacological properties to natural cow bile. It can not only effectively solve the problem of shortage of natural cow bile resources and high cost, but also has significant advantages in quality control.

Research Significance: The promotion of in vitro cultivated cow bile in the treatment of post-traumatic brain injury is expected to provide a more economical and effective treatment option for the recovery of consciousness and cognitive functions of TBI patients. Compared with traditional An Gong Niu Huang Wan, Jian Min Da Peng's An Gong Niu Huang Wan (containing in vitro cultivated cow bile) can not only reduce treatment costs, but also improve the stability and consistency of the quality of the drug. The above clinical research can provide scientific basis for including it in relevant treatment guidelines.

Shortcomings and Innovation Points of Existing Studies: Although An Gong Niu Huang Wan, as a traditional drug for promoting neurological function recovery, has achieved certain effects in some patients, there is a lack of standardized clinical research. The instability of treatment effects in different types of patients has led to the lack of wide recognition from clinical physicians. While in vitro cultivated cow bile is an emerging treatment method, it still lacks sufficient clinical research support. Therefore, this study fills this research gap by comparing the effect of the experimental group (Jian Min Da Peng An Gong Niu Huang Wan group) and the control group (Tong Ren Tang An Gong Niu Huang Wan group) on the recovery of neurological function in post-traumatic brain injury patients, which is highly innovative.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with brain trauma;
2. Age range: 18 - 60 years old (inclusive of 18 and 60);
3. Within three days after injury (for surgical patients, starting from the time of surgery), vital signs are stable (average arterial pressure does not continuously fall below 70 mmHg, no use of vasopressor drugs; no use of invasive or non-invasive ventilators), and the condition is stable (comparison of neurological symptoms and signs at 24-hour intervals and re-examination of CT shows no significant deterioration);
4. GCS score 6 - 12 points (inclusive of 6 and 12), with consciousness disorder;
5. No contraindications for taking artificial or natural rhinoceros bile.

Exclusion Criteria:

1. Have used other arousal-enhancing drugs recently;
2. Patients with consciousness disorders caused by traditional Chinese medicine-induced cold closure of the mind;
3. Patients with open head trauma who have a clear intracranial infection;
4. Patients with severe complications in other organs (such as severe pneumonia, gastrointestinal bleeding, etc.);
5. Patients who have previously suffered from other neurological diseases;
6. Patients with severe acute or chronic diseases in various systems whose conditions have not been effectively controlled and are unstable. This includes, but is not limited to, patients with severe heart diseases such as heart function insufficiency, untreated heart failure, coronary heart disease, severe arrhythmias and other serious cardiac diseases; uncontrolled diabetes, hypertension/low blood pressure, blood system, digestive tract and respiratory system diseases, active autoimmune diseases, etc. Liver and kidney function impairment (liver function: ALT or AST ≥ 2 times the upper limit of normal, total bilirubin > 1.5 times the upper limit of normal; kidney function: Cr > 2 times the upper limit of normal); abnormal coagulation function (PT prolongation > 3 seconds, APTT prolongation > 3 seconds, platelet count < 30 x 109/L). Pregnant and lactating women;
7. Patients who cannot undergo subsequent assessment;
8. Patients considered unsuitable to participate in the trial by the researchers.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
The changes in GCS scores before and after treatment 2 week | 2 week
  We compared the improvement effects of oral administration of Jianmin Dapeng An Gong Niu Huang Wan (containing in vitro cultivated rhinoceros horn) and Tong Ren Tang An Gong Niu Huang Wan (containing natural rhinoceros horn) on the recovery of neurological function in patients with brain trauma after surgery (calculation method: compare the changes in GCS before and after treatment of the two groups, the improvement effect of neurological function = final GCS test score - GCS test score before treatment)

SECONDARY OUTCOMES:
The changes in GCS scores before and after treatment 1 week | 1 week
  We compared the improvement effects of oral administration of Jianmin Dapeng An Gong Niu Huang Wan (containing in vitro cultivated rhinoceros horn) and Tong Ren Tang An Gong Niu Huang Wan (containing natural rhinoceros horn) on the recovery of neurological function in patients with brain trauma after surgery (calculation method: compare the changes in GCS before and after treatment of the two groups, the improvement effect of neurological function = final GCS test score - GCS test score before treatment)
Inflammatory factors: the levels of Inflammatory factors(IL-2, IL-6, WBC, neutrophils, lymphocytes, monocytes, platelets) | 1 week and 2 week
  The levels of inflammatory factors (IL-2, IL-6, WBC, neutrophils, lymphocytes, monocytes, platelets) in brain injury patients one week and two weeks after oral administration of Jianmin Dapeng An Gong Niu Huang Wan (containing in vitro cultivated ox bile) and Tong Ren Tang An Gong Niu Huang Wan (containing natural ox bile) for treatment were compared with those before treatment.
Brain injury indicators: The levels of brain injury indicators (GFAP, NSE, S100-beta) | 1 week and 2 week
  Brain injury indicators: The levels of brain injury indicators (GFAP, NSE, S100-beta) in patients with brain trauma after surgery, one week and two weeks after taking Jianmin Dapeng An Gong Niu Huang Pills (containing in vitro cultivated ox bile) and Tongrentang An Gong Niu Huang Pills (containing natural ox bile) were compared with those before treatment.
Imaging assessment: MRI and CT | 1 week and 2 week
  Imaging assessment: This includes MRI and CT. Observing the recovery of the restoration of normal neural tissue structure in patients with brain trauma after one week and two weeks of oral administration of Jianmin Daopeng Anjungniuhuang Wan (containing in vitro cultivated rhinoceros horn) and Tongrentang Anjungniuhuang Wan (containing natural rhinoceros horn) treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Huaqiu Zhang, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No